CLINICAL TRIAL: NCT00639028
Title: Comparative Study of Two Radiological Modalities, Ultrasonography Versus Stress Radiography, in the Urgent Care and Prognosis of Lateral Ankle Sprains.
Brief Title: Comparative Study of Two Radiological Modalities, Ultrasonography Versus Stress Radiography, in the Urgent Care and Prognosis of Lateral Ankle Sprain (TALOS)
Acronym: TALOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: DCIC 07 02
Record Dates: First submitted 2008-03-11; First posted 2008-03-19 (Estimated); Last update posted 2014-01-23 (Estimated); Status verified 2014-01

CONDITIONS: Lateral Ankle Sprain
Keywords: ankle; diagnosis; sprain; care; injury; stress radiography; ultrasonography
MeSH Terms: conditions — Disease; Sprains and Strains; Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Other): Ankle echography
  Interventions: Other: Ankle echography
- 2 (Other): echography + stress radiography
  Interventions: Other: Ankle echography + stress radiography
- 3 (Other): stress radiography
  Interventions: Other: stress radiography

INTERVENTIONS:
Other: Ankle echography — Ankle echography
  Arms: 1
Other: Ankle echography + stress radiography — Ankle echography + stress radiography
  Arms: 2
Other: stress radiography — ankle stress radiography
  Arms: 3

SUMMARY:
The aim of our study is to determine the most efficient radiologic examination to assess the ankle sprain seriousness and so improve the therapeutic care.

DETAILED DESCRIPTION:
The lateral ankle sprain is the most frequent purpose of consultation in emergency traumatology of the locomotive system.

If the ankle sprain is neglected or badly cared, it can induce a recurrence or several complications particularly functional ones. So a gravity diagnosis is necessary in order to choose the most accurate treatment.

Considering the difficulty of the clinical estimation, additional examinations aim to support the positive diagnosis, to clarify the gravity and to dismiss differential diagnosis.

Thus we suggest to evaluate three strategies in order to get a gravity diagnosis, make a better choice of treatment and so decrease the long-term functional complications : instability and recurrence.

The patients are randomly separated into three groups of 130 people. All the patients have a radiography and then, according to their group, they have either an ultrasonography or an ultrasonography and a stress radiography or only a stress radiography. The patients are followed up during two years by sending two questionnaires (CAIT and LEFS) at one and two years. The functional scores of these questionnaires assess and compare the functional complications for each group. Thus the radiologic examinations can be assessed in term of prognosis.

ELIGIBILITY:
Inclusion Criteria:

* Lateral ankle sprain.
* Sprain occurred for less than 48 hours.
* Age between 18 and 55.
* Person affiliated at the Social Security.

Exclusion Criteria:

* Recurrent lateral ankle sprain occurred for less than 2 years and diagnosed by a doctor.
* Bilateral sprain, medio-tarsal sprain, syndesmosis sprain, subtalar sprain.
* Tendinous luxation (fibular, posterior tibial).
* Homolateral ankle fracture occurred for less than 2 years.
* Cuboid fracture, external tubercle of astragalus fracture, calcaneum fracture, fracture of the talus extremity, base of the fifth metatarsal bone fracture.
* Tearing of internal malleolus, tearing of astragalus posterior tubercle.
* Osteochondral lesions of the astragalus dome.
* Probable difficulty to follow up the patient.
* Patient taking anticoagulant.
* Pregnant woman, parturient, breast-feeding mother.
* Person deprived of freedom after a judicial or an administrative decision, person with legal protection measure.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 390 (Estimated)
Dates: Start 2007-11; Primary Completion 2013-12 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Residual ankle instability evaluated using the Cumberland Ankle Instability Tool (CAIT) | at one year

SECONDARY OUTCOMES:
Lower Extremity Functional Squale (LEFS) Score | at one year
Lower Extremity Functional Squale (LEFS) Score | at two years
Baecke Physical Activity Questionnaire Score | at the clinical examination
Cumberland Ankle Instability Tool (CAIT) Score | at two years
Number of lesions in the group echography/stress radiography versus in the group echography. | at the clinical examination

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Jacques Banihachemi, Principal Investigator — University Hospital, Grenoble
Locations (1):
- Emergency department - University Hospital of Grenoble South, Grenoble, France

REFERENCES:
- [Background] Picard F, Tourne Y, Montbarbon E, Saragaglia D. [Ankle trauma. Diagnostic orientation]. Rev Prat. 1995 Nov 15;45(18):2335-42. No abstract available. French. PMID 8578138
- [Background] Braun BL. Effects of ankle sprain in a general clinic population 6 to 18 months after medical evaluation. Arch Fam Med. 1999 Mar-Apr;8(2):143-8. doi: 10.1001/archfami.8.2.143. PMID 10101985
- [Background] Brasseur JL, Tardieu M. [Accurate use of imaging in ankle sprain]. JBR-BTR. 1999 Apr;82(2):63-8. French. PMID 10874392
- [Background] Raatikainen T, Putkonen M, Puranen J. Arthrography, clinical examination, and stress radiograph in the diagnosis of acute injury to the lateral ligaments of the ankle. Am J Sports Med. 1992 Jan-Feb;20(1):2-6. doi: 10.1177/036354659202000102. PMID 1554068
- [Background] Brasseur JL, Morvan G, Godoc B. [Dynamic ultrasonography]. J Radiol. 2005 Dec;86(12 Pt 2):1904-10. doi: 10.1016/s0221-0363(05)81544-6. French. PMID 16308555
- [Background] Hiller CE, Refshauge KM, Bundy AC, Herbert RD, Kilbreath SL. The Cumberland ankle instability tool: a report of validity and reliability testing. Arch Phys Med Rehabil. 2006 Sep;87(9):1235-41. doi: 10.1016/j.apmr.2006.05.022. PMID 16935061